CLINICAL TRIAL: NCT02818530
Title: Correlation Between Intraocular Pressure Measurement by Tomometer and Anterior Chamber Depth Measurement by Ultrasound in Steep Trendelenberg Position During Robotic Assisted Surgery
Brief Title: Correlation Between Intraocular Pressure Measurement by Tomometer and Anterior Chamber Depth Measurement by Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Two patients developed corneal laceration and hence study re-reviewed by IEC and decided to terminate the study prematurely
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Sohan Lal Solanki, Assistant Professor, Department of Anesthesiology, Critical Care and Pain, Tata Memorial Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PN 1690
Record Dates: First submitted 2016-06-18; First posted 2016-06-29 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Urological Cancer; Gastrointestinal Cancer; Malignant Female Reproductive System Neoplasm
MeSH Terms: conditions — Urologic Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOP by tomoneter and ultrasound (Experimental): Intraocular pressure will be measured by electronic tomometer (tonopen) at different point of time after induction of anaesthesia in patients undergoing robotic assisted surgery under steep Trendelenberg position. Anterior chamber depth will be measured by ultrasound at the same time intervals.
  Interventions: Device: IOP by tonometer; Device: Anterior chamber depth measurement by ultrasound

INTERVENTIONS:
Device: IOP by tonometer — Electronic tonometer will be used as gold standard for intraocular pressure measurement in supine position after induction of anaesthesia and every 2 hours intraoperatively and at end of surgery.
Device: Anterior chamber depth measurement by ultrasound — Anterior chamber depth will be measured by ultrasound in supine position after induction of anaesthesia and every 2 hours intraoperatively and at end of surgery.

SUMMARY:
Intra ocular pressure (IOP) may theoretically increase due to steep Trendelenberg position and studies showed that IOP reaches peak levels after steep Trendelenberg position on an average of 13 mmHg higher than preanesthesia induction values. Major determinants of IOP are aqueous humor flow, choroidal blood volume, central venous pressure and extra ocular muscle tone.

Hassen GW et al measured anterior chamber depth in 2 patients with glaucoma and compared the anterior chamber depth (ACD) with the intraocular pressure measured by tonometer. They concluded that bedside ultrasound could be useful in evaluating patient with suspected increased IOP, who are unable to open their eyes.

DETAILED DESCRIPTION:
Intra ocular pressure (IOP) may theoretically increase due to steep Trendelenberg position and studies showed that IOP reaches peak levels after steep Trendelenberg position on an average of 13 mmHg higher than preanesthesia induction values. Major determinants of IOP are aqueous humor flow, choroidal blood volume, central venous pressure and extra ocular muscle tone. During the robotic surgery there are two theories explaining the increase of IOP, first, gravitational forces increase central venous pressure which in turn affect orbital venous pressure and increase IOP. Second, intraperitoneal carbon dioxide causes increased choroidal blood volume which may result in IOP increase. One study reported that low end tidal carbon dioxide was a significant predictor of the IOP increase. Continuous absorption of carbon dioxide from peritoneum and increased pressure on diaphragm results in lower delivered tidal volumes and subsequently increased arterial carbon dioxide levels leading to increased choroidal blood flow and increased IOP.

Hassen GW et al measured anterior chamber depth in 2 patients with glaucoma and compared the anterior chamber depth (ACD) with the intraocular pressure measured by tonometer. They concluded that bedside ultrasound could be useful in evaluating patient with suspected increased IOP, who are unable to open their eyes. It can also be used for serial examination and follow-up of treatment success. They also mentioned that, it is necessary to conduct a prospective study with a larger sample size, to evaluate if there is agreement between measurements using a tonometer and measurements of the ACD using ultrasound. In addition, it is essential to determine the cut off normal ACD for evaluation of IOP.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-III
2. Urological cancer patients under going robotic assisted surgeries.
3. Gastrointestinal cancer patients under going robotic assisted surgeries,
4. Gynecological cancer patients under going robotic assisted surgeries,

Exclusion Criteria:

1. ASA class IV and above
2. Patients with a history of glaucoma.
3. Patients with corneal disease, retinal vascular disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure measured by tonometer | Just after induction of anesthesia, every 2 hours during surgery and immediately after surgery
  Intra operative recordings of IOP will be after induction and thereafter will be measured every 2 hours and at the end of surgery.
Changes in anterior chamber depth measured by ultrasound. | Just after induction of anesthesia, every 2 hours during surgery and immediately after surgery
  Intra operative recordings of anterior chamber depth will be measured after induction of anaesthesia, every 2 hours intraoperatively and at end of surgery.

SECONDARY OUTCOMES:
Time dependent changes in IOP during prolonged steep Trendelenberg position. | Just after induction of anesthesia, every 2 hours during surgery and immediately after surgery
Time dependent changes in anterior chamber depth during prolonged trendelenberg position. | Just after induction of anesthesia, every 2 hours during surgery and immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sohan L Solanki, MD, Principal Investigator — Tata Memorial Centre
Locations (1):
- Sohan Lal solanki, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided